CLINICAL TRIAL: NCT06372821
Title: A Randomized, Participant & Investigator Blinded, Placebo-Controlled Study to Evaluate the Ability of Intrathecally Administered NIO752 to Lower CSF Total Tau Synthesis in Participants With AD Measured by Stable Isotope Labelling Kinetics
Brief Title: A Trial Evaluating the Effect of NIO752 on Tau Synthesis Measured by a Process Known as SILK
Acronym: NIO-SILK
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Washington University School of Medicine (Other); University of Washington (Other); Alzheimer's Association (Other); Sigrid Rausing Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 158160
Record Dates: First submitted 2024-03-13; First posted 2024-04-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Autosomal Dominant Alzheimer Disease Due to Mutation of Presenilin 1 (Disorder); Autosomal Dominant Alzheimer Disease Due to Mutation of Presenilin 2 (Disorder); Autosomal Dominant Alzheimer Disease Due to Mutation of Amyloid Precursor Protein (Disorder)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NIO752 (Experimental): Intrathecal administration.
  Interventions: Drug: NIO752
- Saline (Placebo Comparator): 10mL of saline (placebo) is administered intrathecally.
  Interventions: Drug: NIO752; Other: Placebo

INTERVENTIONS:
Drug: NIO752 — Antisense oligonucleotide
Other: Placebo — Saline
  Arms: Saline

SUMMARY:
This study will assess if drug (NIO752) reduces production of a protein, tau, by the brain. Normally tau maintains the internal skeleton of nerve cells. In Alzheimer's disease (AD) it builds up in the brain, causing damage. Abnormal tau proteins cling to each other forming 'tangles' inside nerve cells, which interfere with how the nerve cells work, and eventually die. This is what causes the symptoms of dementia. It is thought that NIO752 reduces production of tau.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide signed informed consent.
2. Between 21 to 80 years old (inclusive).
3. A diagnosis of mild or moderate Alzheimer's disease by a Clinical Dementia Rating score of 0.5 to 2, where the investigator believes they will be able to complete the study.
4. A history of cerebrospinal fluid, Positron Emission Topography (PET), or blood-based biomarkers supporting the diagnosis of Alzheimer's disease, or symptomatic approved presenilin (PSEN) or amyloid precursor protein (APP) mutation carriers. If blood biomarkers are equivocal then amyloid status can be confirmed using cerebrospinal fluid.
5. Fluency in English
6. Participant has a reliable study partner or caregiver
7. Able to undergo lumbar punctures, magnetic resonance imaging (MRI), cerebrospinal fluid draws, and blood draws.
8. Individuals will be willing to consent for their biological samples and personal data to be shared with the commercial partner (Novartis)

Exclusion Criteria:

1. Live in a skilled nursing facility or dementia care facility.
2. Any clinically significant laboratory abnormality
3. Attempted suicide, suicidal ideation with a plan that required hospital admission within 12 months prior to Screening
4. Any previous use of experimental therapy within 180 days or 5 half-lives prior to Day 1, whichever is greater.
5. Any previous use of MAPT antisense oligonucleotides (ASO) or any other ASO or other gene therapy meant as treatment for Alzheimer's disease.
6. History of hypersensitivity to any of the study treatments or its excipients or to drugs of similar chemical classes.
7. Any condition that increases risk of meningitis unless participant is receiving appropriate prophylactic treatment.
8. Current medical or non-Alzheimer's disease neurological condition that might impact cognition or performance on cognitive assessments
9. Have any other conditions which, in the opinion of the investigator, would make the participant unsuitable for inclusion or could interfere with the patient participating in or completing the study.
10. Unlikely to cooperate in the study; not able to attend scheduled examinations and visits; or not able to follow study instructions per the judgement of the investigator.
11. Current alcohol (>14 units per week) or current cannabis use; or history of alcohol or drug abuse or dependence (except nicotine dependence) within 2-years before the screening visit.
12. Treatment with immunosuppressants, antipsychotics, lithium, neuroleptics, dopaminergic agonists, L-dopa, or monoamine oxidase inhibitors at the time of screening. Current use of medications, other than cholinesterase inhibitors and/or memantine, that could alter cognition, as determined by the Investigator. If patients are taking cholinesterase inhibitors and/or memantine at screening, the dose must have been stable within 12-weeks prior to screening and must remain stable during the duration of the study.
13. Unable to undergo MRI due to for example claustrophobia, or presents absolute contraindications to MRI (e.g., metallic implants, metallic foreign bodies, pacemaker, defibrillator).
14. Significant signs of major cerebrovascular disease
15. Sexually active males, unless they agree to use a condom during intercourse from the time of consent until a minimum of 15 weeks after treatment.
16. Breast feeding women, pregnant women, and females of reproductive potential unless they use highly effective contraception methods, as specified in the protocol.
17. Patients on regular anticoagulants or anti-platelets that would preclude lumbar puncture are not eligible to participate
18. Seropositive for human immunodeficiency virus (HIV), Hepatitis B or hepatitis C.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Tau synthesis rate inhibition in individuals with sporadic AD and ADAD | Day 23
  Tau synthesis rate calculated using tracer to tracee ratio of tau specific peptide calculated on day 20 post leucine administration in individuals with sporadic and ADAD (analyzed collectively) receiving intrathecal NIO752 compared to placebo.

SECONDARY OUTCOMES:
Compare efficacy of knockdown of tau production in sporadic AD and ADAD by measuring the synthesis rate of tau by determining the ratio of labelled to unlabeled tau (tracer to tracee ratio) in serial cerebrospinal fluid samples. | Day 23
Number of participants with adverse events [safety and tolerability] | Day 0 to Day 145
Comparison of number of Adverse Events reported between participants receiving one dose of NIO752 versus those receiving two doses of NIO752. | Day 0 to Day 145
  Compare safety between 1 and 2 doses.
Compare rates of tau synthesis and clearance in sporadic AD and ADAD | Day 23
Determine CSF tau concentration to tau production relationships in humans | 120 days

CONTACTS AND LOCATIONS:
Locations (2):
- Washington University in St. Louis, St Louis, Missouri, United States
- University College London Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No